CLINICAL TRIAL: NCT04182724
Title: Camrelizumab, Apatinib and Nab-paclitaxel as Second-line Treatment in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Camrelizumab GC
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — camrelizumab; apatinib; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab, Apatinib and Nab-paclitaxel (Experimental): Camrelizumab was administered 200mg iv every 2 weeks, Apatinib 250 mg p.o. qd Nab-paclitaxel 125 mg/m2, 150 mg/m2, 175 mg/m2 or 200 mg/m2, iv. q2w
  Interventions: Drug: Camrelizumab, Apatinib and Nab-paclitaxel

INTERVENTIONS:
Drug: Camrelizumab, Apatinib and Nab-paclitaxel — Camrelizumab was administered 200mg iv every 2 weeks, Apatinib was administered 250 mg p.o. qd Nab-paclitaxel was administered 125 mg/m2, 150 mg/m2, 175 mg/m2 or 200 mg/m2, iv. q2w

SUMMARY:
This is a Phase I/II , Open-label , Investigator-initiated Trail of Camrelizumab (an Anti-PD-1 Inhibitor), Apatinib (VEGFR2 Inhibitor) and Nab-paclitaxel as Second-line Treatment in Advanced Gastric Cancer The study was designed in two stages, the first stage was the tolerance observation stage, and the second stage was the curative effect expansion stage.

The first part of the study is the Dose-finding Phase designed to establish the safety of Camrelizumab, Apatinib and Nab-paclitaxel at different dose Levels(125 mg/m2, iv. q2w, 150 mg/m2, iv. q2w, 175 mg/m2, iv. q2w or 200 mg/m2, iv. q2w). The second part of the study is the Expansion Phase designed to generate additional clinical data at specified doses .

This study aims to evaluate the safety and efficacy of Camrelizumab, Apatinib and Nab-paclitaxel in the Second-line treatment of advanced Gastric Cancer.

DETAILED DESCRIPTION:
This trial investigated the safety and efficacy of Camrelizumab, Apatinib and Nab-paclitaxel as Second-line Treatment in Advanced Gastric Cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: more than 18 years old, male or female;
* 2.Pathologically diagnosed with advanced gastric cancer (including adenocarcinoma of the gastroesophageal junction) with measurable metastases outside the stomach (measuring ≥ 10mm on spiral computed tomography(CT) scan, satisfying the criteria in Response Evaluation Criteria In Solid Tumors (RECIST) 1.1);
* 3.Failure of prior therapy (during or after treatment) in patients who have received at first line chemotherapy regimens(platinum - based regimens);
* 4.Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1;
* 5.Major organ function has to meet the following criteria: Hemoglobin (HB) ≥ 80g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 90 × 109 / L, ALT and AST ≤ 2.5 × ULN, liver metastases, the ALT and AST≤5 × ULN, Bilirubin ≤ 1.5 times the upper limit of normal (ULN), Serum creatinine ≤ 1.5 times the upper limit of normal (ULN),
* 6.An expected survival of ≥ 3 months;
* 7.Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 12 week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 12 week post the last administration of study drug;
* 8.Patient has to voluntarily join the study and sign the Informed Consent Form for the study.

Exclusion Criteria:

* 1．Other malignancies have been diagnosed within 5 years prior to the first use of the study drug, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or cervical and/or breast cancer in situ which have been effectively treated;
* 2．Subjects are using immunosuppressive agents.
* 3．Confirmed that Camrelizumab, Apatinib, Nab-paclitaxel and/or its accessories allergy;
* 4．Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
* 5．Peripheral neuropathy >1 grade;
* 6．Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than Class Ⅰ; Ⅰ-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class Ⅰ cardiac dysfunction; Patients with positive urinary protein;
* 7．Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 2 months;unresected primary lesion in stomach with positive fecal occult blood test (+), ulcerated gastric carcinoma with massive alimentary tract bleeding risk judged by PIs based on gastric endoscopy result;
* 8．Abnormal Coagulation (INR>1.5、APTT>1.5 UNL), with tendency of bleed;
* 9．Associated with CNS (central nervous system) metastases;
* 10．Pregnant or lactating women;
* 11．With psychotropic drug abuse history and can't get rid of or mental disorder patients;
* 12．Participated in other clinical trials within 4 weeks;
* 13．Any other condition that might place the patient at undue risk or preclude a patient from completing the study;
* 14．Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-05-12 (Estimated); Study Completion 2022-05-12 (Estimated)

PRIMARY OUTCOMES:
MTD /DLT (phase I) | Within four weeks after administration
  Maximum Tolerated Dose/Dose Limiting Toxicity
ORR(phase II) | from the first drug administration up to two years
  Overall Response Rate

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (phase I/II) | from the first drug administration to within 90 days for the last drug dose
  adverse events/serious adverse events
PFS(phase I/II) | from the first drug administration up to two years
  Progression-Free-Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gou M, Zhang Y, Wang Z, Qian N, Dai G. PD-1 inhibitor combined with albumin paclitaxel and apatinib as second-line treatment for patients with metastatic gastric cancer: a single-center, single-arm, phase II study. Invest New Drugs. 2024 Apr;42(2):171-178. doi: 10.1007/s10637-024-01425-3. Epub 2024 Feb 12. PMID 38347177